CLINICAL TRIAL: NCT00488462
Title: Non-Pneumatic Anti-Shock Garment for Obstetrical Hemorrhage: Zambia and Zimbabwe
Acronym: NASG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Bill and Melinda Gates Foundation (Other); University of Zambia (Other); University of Zimbabwe (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HD053129-01A1 (NIH); 5R01HD053129-03 (NIH)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Hypovolemic Shock; Hemorrhage
Keywords: obstetric hemorrhage; hypovolemic shock; non-pneumatic anti-shock garment; safe motherhood; maternal mortality; maternal morbidity
MeSH Terms: conditions — Shock; Hemorrhage; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Clinics will collect data on patients experiencing shock due to obstetrical hemorrhage. In the control arm, half of the study clinics will not use the NASG but the NASG will be available at the referral hospital for patients transported there.
- Intervention (Other): Clinics will collect data on patients experiencing shock due to obstetrical hemorrhage. In the intervention arm, half of the study clinics will use the NASG on patients before transporting to the referral hospital.
  Interventions: Device: non-pneumatic anti-shock garment

INTERVENTIONS:
Device: non-pneumatic anti-shock garment — In the intervention arm, half of the study clinics will use the NASG when a patient meets the study criteria.
  Other Names: NASG; Anti-Shock Garment; Manufactured by Zoex; Life Wrap
  Arms: Intervention

SUMMARY:
This trial will address the question of whether early application of the Non-pneumatic Anti-Shock Garment (NASG) at the Satellite Health Facility (SHF) level before transport to a Referral Hospital (RH) will decrease maternal mortality and morbidity. The available evidence indicates that the NASG substantially decreases blood loss, but there is no evidence that its application will reduce extreme adverse outcomes. It is also not known if possible side effects associated with NASG use might outweigh potential benefits. This study would rigorously test the effectiveness of the NASG using an experimental design with adequate power to detect statistically significant decreases in morbidity and mortality.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial to examine the effects of NASG application as a first-aid device at the SHFs before transfer to Referral Hospitals (RHs).

The first step will include start-up activities and formative data collection, including facility staff training in data collection, how to collect blood in the closed-end blood collection drape, and in an evidence-based standardized clinical protocol for obstetric hemorrhage prevention and hemorrhage and shock management. Next will be a period of baseline data collection at the RHs and SHFs, during which clinical and demographic data will be collected from women diagnosed with obstetric hemorrhage and shock. After this baseline data collection period, we will introduce the study intervention, initially at the RHs and then at SHFs.

The intervention will include: review of study protocol differences between baseline and the NASG-intervention phases, provision of the NASG, detailed training on the use of NASG for health care providers and staff, as well as on-site support and supervision for use of the NASG. After the RH providers are fully trained and have become proficient in NASG use, SHFs will be randomized into 19 intervention and 19 control facilities. Intervention SHFs will receive the NASG training described above, while control SHFs will receive a refresher training on the topics included in the baseline training.

The final step will be three years of NASG-intervention data collection at the RHs and the SHFs on women diagnosed with obstetric hemorrhage and shock on the same outcomes collected in the baseline period. A total of approximately 2,340 women from the SHFs will be included in the NASG-intervention data collection phase of the cluster randomized trial: 1,170 women in the intervention group and 1,170 women in the control group.

ELIGIBILITY:
To participate in these study activities, women must be willing and able to participate, be able to sign or mark a consent form, and speak one of the languages into which the consent form has been translated, including English, Nyanja, and Bemba in Zambia, and English, Shona and Ndebele in Zimbabwe.

Inclusion Criteria:

* Women who are pregnant or postpartum and experiencing obstetric hemorrhage with 2 of the following 3:

blood loss > 500 mL (at SHF, 1000 mL at RH) SBP <100 mm Hg pulse >100 bpm

Exclusion Criteria:

* Absolute exclusion criteria include: current viable third trimester intrauterine pregnancy that can be delivered in the next 20 minutes after hemorrhage begins and/or current bleeding sites above the diaphragm. Relative exclusion criteria include: a history or current clinical evidence of mitral stenosis or congestive heart failure (CHF). These must be relative contraindications that will be assessed at the time of hemorrhage and clinical judgment will need to be utilized to evaluate each case individually. Thus if the patient can be transported and delivered rapidly and is suspected or known to have valvular heart disease, she will be excluded from the study. In other cases, depending on the severity of the hemorrhage, if the patient is dyspneic in the NASG, at the SHF level, the NASG will be loosened, if that does not result in relief, the NASG will be removed. If the patients at the RH have decreasing oxygen saturation levels as demonstrated by pulse oximeter, the NASG will be loosened, if that does not result in relief, the NASG will be removed.

Women suffering obstetric hemorrhage and hypovolemic shock who have no detectable vital signs (non palpable pulse and BP) at the time of their arrival at the RH are ineligible for enrolment in the study ("non-resuscitable") if: 1) the woman does not respond to resuscitation attempts after 30 minutes and 2) more than three hours have elapsed between the start of hemorrhage and the beginning of her treatment. (As this is a clinical intervention of a potentially life saving device, the study clinicians should try the NASG on any patient if they feel it may resuscitate her; however, if the woman meets the criteria above they are ineligible for having their data entered into the study.)

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2007-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Frequency of mortalities and frequency of severe morbidities combined as extreme adverse outcomes | during hospital stay

SECONDARY OUTCOMES:
Mean amount of blood loss in mL , frequency of emergency hysterectomy, time to recovery from shock. | during hospital stay
  Blood loss as measured by the blood collection drape at the RH or pad between SHF and RH.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Miller, CNM, PhD, Principal Investigator — University of California, San Francisco; Elizabeth Butrick, MPH, MSW, Study Director — University of California, San Francisco; Thulani Magwali, OBGYN, Principal Investigator — University of Zimbabwe Hospital, Harare, Zimbabwe (UZ); Gricelia Mkumba, OBGYN, Principal Investigator — University Teaching Hospital, Lusaka Zambia (UTH)
Locations (5):
- Zambia (3):
  - Kitwe Central Hospital, Kitwe, Copperbelt
  - Ndola Central Hospital, Ndola, Copperbelt
  - University Teaching Hospital (UTH), Lusaka
- Zimbabwe (2):
  - Harare Hospital, Harare
  - Parienyatwa Group of Hospitals, Harare

REFERENCES:
- [Background] Miller S, Hamza S, Bray EH, Lester F, Nada K, Gibson R, Fathalla M, Mourad M, Fathy A, Turan JM, Dau KQ, Nasshar I, Elshair I, Hensleigh P. First aid for obstetric haemorrhage: the pilot study of the non-pneumatic anti-shock garment in Egypt. BJOG. 2006 Apr;113(4):424-9. doi: 10.1111/j.1471-0528.2006.00873.x. PMID 16553654
- [Background] Brees C, Hensleigh PA, Miller S, Pelligra R. A non-inflatable anti-shock garment for obstetric hemorrhage. Int J Gynaecol Obstet. 2004 Nov;87(2):119-24. doi: 10.1016/j.ijgo.2004.07.014. PMID 15491555
- [Background] Miller S, Hensleigh P. Non-pneumatic Anti-shock Garment for Obstetric Hemorrhage. Chapter 14 in: (eds) B-Lynch, C, Keith, L, LaLonde, A, Karoshi, M. An International Federation of Obstetrics and Gynecology (FIGO) Book Postpartum Hemorrhage: New Thoughts, New Approaches. London, UK: Sapiens Publications; 2006. p. 136-46.
- [Background] Miller S, Ojengbede A, Turan JM, Ojengbede O, Butrick E, Hensleigh P. Anti-Shock Garments for Obstetric Hemorrhage. Current Women's Health Reviews. 2007;3(1):3-11.
- [Background] Miller S, Turan JM, Dau K, Fathalla M, Mourad M, Sutherland T, Hamza S, Lester F, Gibson EB, Gipson R, Nada K, Hensleigh P. Use of the non-pneumatic anti-shock garment (NASG) to reduce blood loss and time to recovery from shock for women with obstetric haemorrhage in Egypt. Glob Public Health. 2007;2(2):110-24. doi: 10.1080/17441690601012536. PMID 19280394
- [Background] Miller S, Turan JM, Ojengbede A, Ojengbede O, Fathalla M, Morhason-Bello IO, Youssif MM, Galandanci H, Hamza S, Awwal M, Akinwuntan A, Mohammed AI, McDonough L, Dau K, Butrick E, Hensleigh P. The pilot study of the non-pneumatic anti-shock garment (NASG) in women with severe obstetric hemorrhage: Combined results from Egypt and Nigeria. Int J Gynaecol Obstet. 2006 Nov;94 Suppl 2:S154-S156. doi: 10.1016/S0020-7292(06)60022-2. No abstract available. PMID 29644686
- [Background] Miller S, Martin HB, Morris JL. Anti-shock garment in postpartum haemorrhage. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):1057-74. doi: 10.1016/j.bpobgyn.2008.08.008. Epub 2008 Sep 20. PMID 18805742
- [Background] Miller S, Ojengbede O, Turan JM, Morhason-Bello IO, Martin HB, Nsima D. A comparative study of the non-pneumatic anti-shock garment for the treatment of obstetric hemorrhage in Nigeria. Int J Gynaecol Obstet. 2009 Nov;107(2):121-5. doi: 10.1016/j.ijgo.2009.06.005. Epub 2009 Jul 22. PMID 19628207
- [Background] Miller S, Fathalla MM, Youssif MM, Turan J, Camlin C, Al-Hussaini TK, Butrick E, Meyer C. A comparative study of the non-pneumatic anti-shock garment for the treatment of obstetric hemorrhage in Egypt. Int J Gynaecol Obstet. 2010 Apr;109(1):20-4. doi: 10.1016/j.ijgo.2009.11.016. Epub 2010 Jan 22. PMID 20096836
- [Background] Mourad-Youssif M, Ojengbede OA, Meyer CD, Fathalla M, Morhason-Bello IO, Galadanci H, Camlin C, Nsima D, Al Hussaini T, Butrick E, Miller S. Can the Non-pneumatic Anti-Shock Garment (NASG) reduce adverse maternal outcomes from postpartum hemorrhage? Evidence from Egypt and Nigeria. Reprod Health. 2010 Sep 1;7:24. doi: 10.1186/1742-4755-7-24. PMID 20809942
- [Background] Miller S, Fathalla MM, Ojengbede OA, Camlin C, Mourad-Youssif M, Morhason-Bello IO, Galadanci H, Nsima D, Butrick E, Al Hussaini T, Turan J, Meyer C, Martin H, Mohammed AI. Obstetric hemorrhage and shock management: using the low technology Non-pneumatic Anti-Shock Garment in Nigerian and Egyptian tertiary care facilities. BMC Pregnancy Childbirth. 2010 Oct 18;10:64. doi: 10.1186/1471-2393-10-64. PMID 20955600
- [Background] Ojengbede OA, Morhason-Bello IO, Galadanci H, Meyer C, Nsima D, Camlin C, Butrick E, Miller S. Assessing the role of the non-pneumatic anti-shock garment in reducing mortality from postpartum hemorrhage in Nigeria. Gynecol Obstet Invest. 2011;71(1):66-72. doi: 10.1159/000316053. Epub 2010 Dec 15. PMID 21160197
- [Background] Turan J, Ojengbede O, Fathalla M, Mourad-Youssif M, Morhason-Bello IO, Nsima D, Morris J, Butrick E, Martin H, Camlin C, Miller S. Positive effects of the non-pneumatic anti-shock garment on delays in accessing care for postpartum and postabortion hemorrhage in Egypt and Nigeria. J Womens Health (Larchmt). 2011 Jan;20(1):91-8. doi: 10.1089/jwh.2010.2081. Epub 2010 Dec 29. PMID 21190486
- [Background] Fathalla MM, Youssif MM, Meyer C, Camlin C, Turan J, Morris J, Butrick E, Miller S. Nonatonic obstetric haemorrhage: effectiveness of the nonpneumatic antishock garment in egypt. ISRN Obstet Gynecol. 2011;2011:179349. doi: 10.5402/2011/179349. Epub 2011 Aug 10. PMID 21845226
- [Background] Morris, J., Meyer, C., Fathalla, MF, Youssif, MM, Al-Hussaini, TK, Camlin, C., Miller, S. Treating Uterine Atony with the NASG in Egypt. African Journal of Midwifery and Women's Health 5(1):37-42, 2011
- [Background] Ojengbede, O., Galadanci, H., Morhason-Bello, IO, Nsima, D., Camlin, C., Morris, J., Butrick, E., Meyer, C., Mohammed, AI, Miller, S. The Non-pneumatic Anti-Shock Garment for Postpartum Haemorrhage in Nigeria. African Journal of Midwifery and Women's Health 5(3):135-9, 2011
- [Background] Lester F, Stenson A, Meyer C, Morris J, Vargas J, Miller S. Impact of the Non-pneumatic Antishock Garment on pelvic blood flow in healthy postpartum women. Am J Obstet Gynecol. 2011 May;204(5):409.e1-5. doi: 10.1016/j.ajog.2010.12.054. Epub 2011 Mar 24. PMID 21439543
- [Background] Stenson, A., Lester, F., Meyer, C., Morris, J., Vargas, V., Miller, S. The Non-pneumatic Anti-Shock Garment: How Applier Strength and Body Mass Index Affect Pressure. International Journal of Gynecology and Obstetrics, 2011; 5:33-37
- [Background] Kausar F, Morris JL, Fathalla M, Ojengbede O, Fabamwo A, Mourad-Youssif M, Morhason-Bello IO, Galadanci H, Nsima D, Butrick E, Miller S. Nurses in low resource settings save mothers' lives with non-pneumatic anti-shock garment. MCN Am J Matern Child Nurs. 2012 Sep;37(5):308-16. doi: 10.1097/NMC.0b013e318252bb7d. PMID 22895203
- [Derived] Miller S, Bergel EF, El Ayadi AM, Gibbons L, Butrick EA, Magwali T, Mkumba G, Kaseba C, Huong NT, Geissler JD, Merialdi M. Non-pneumatic anti-shock garment (NASG), a first-aid device to decrease maternal mortality from obstetric hemorrhage: a cluster randomized trial. PLoS One. 2013 Oct 23;8(10):e76477. doi: 10.1371/journal.pone.0076477. eCollection 2013. PMID 24194839
- See also: Information and updates on current trials using the Life Wrap (NASG) for obstetric hemorrhage in low resource settings. — http://www.lifewrap.org